CLINICAL TRIAL: NCT04327648
Title: A Clinical Study to Explore the Effect and Mechanism of Social Interaction on Autism Spectrum Disorder Children: a Randomized Double-blinded Clinical Trial
Brief Title: Effect and Mechanism of Social Interaction Treatment on ASD Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XH-20-004
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: ASD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social interaction treatment (Active Comparator): During the treatment days, children in social interaction treatment group will have 30min social interaction each day for 3 months. ASD children are followed up closely.
  Interventions: Device: Social interaction treatment
- Neuronal cognition treatment (Sham Comparator): Children in neuronal cognition treatment group will experienced neural cognition training 30min each day for 3 months. ASD children are followed up closely.
  Interventions: Device: Neuronal cognition treatment
- Routine treatment (Other): Children in routine treatment group will keep the same initial treatment. ASD children are followed up closely.
  Interventions: Other: Routine treatment

INTERVENTIONS:
Device: Social interaction treatment — Children in social interaction treatment group will have 30min social interaction each day for 3 months.
  Arms: Social interaction treatment
Device: Neuronal cognition treatment — Children in neuronal cognition treatment group will experienced neural cognition training 30min each day for 3 months.
  Arms: Neuronal cognition treatment
Other: Routine treatment — Children in routine treatment group will keep the same initial treatment.
  Arms: Routine treatment

SUMMARY:
Current study try to find out whether social interaction treatment is effective for ASD children. ASD children will be divided into three groups, social interaction treatment group, neuronal cognition treatment and routine treatment group. Based on excited recognition training treatment effect on the core symptom of ADHD by tablet computer, the investigators propose that tablet computer social interaction treatment may induce a significant improvement in ameliorating the social disorder of ASD.

DETAILED DESCRIPTION:
Appropriate and effective treatment coupled with home training can help ASD children restore the ability of language, behavior and learning. However, there is no suitable and effective behavior intervention for home training yet. Current study try a 3 months' randomized double-blinded clinical trial to find out whether tablet computer social interaction treatment at home is effective for ASD children. 90 3-6 years old ASD children will be included and divided into three groups, social interaction treatment group, neuronal cognition treatment and routine treatment group respectively. During the treatment days, children in social interaction treatment group will have 30min social interaction each day for 3 months. Children in neuronal cognition treatment group will experienced neural cognition training 30min each day for 3 months. Children in routine treatment group will keep the same initial treatment. All ASD children are followed up closely. The primary observed indicator is the score of Childhood Autism Rating Scale (CARS) at the inclusion, one month and 3 month after treatment to evaluate the effect of tablet computer social interaction treatment on ASD children.

ELIGIBILITY:
Inclusion criteria：

* Patients diagnosed with ASD. Diagnostic criteria: diagnosed by pediatric psychiatrists in accordance with the criteria in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V), Autism Diagnostic Observation Schedule (ADOS) and Autism Diagnostic Interview-Revised (ADI-R)
* CARS ≥ 34
* Agree to sign the informed consent

Exclusion criteria：

* Children with abnormal gene and chromosome
* Children with neurodevelopmental diseases (like epilepsy, schizophrenia)
* Children with severe sense perception disorder
* Children with weight over 20kg, with electronic metal products in body unsuited for magnetic resonance imaging

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale, (CARS) | The baseline and 3 months after treatment
  CARS is a behaviour-rating scale used to assess the presence and severity of the symptoms of autism spectrum disorder(ASD), with scores ranging from 15 to 60 and high scores indicating severe symptoms. Change of the CARS from baseline to 3 months after treatment to evaluate the effect of tablet computer social interaction treatment on ASD children.

SECONDARY OUTCOMES:
Social responsiveness scale, (SRS) | The baseline and 3 months after treatment
  SRS is a questionnaire used to assess the presence and severity of social impairment, with high scores indicating severe symptoms. Change of the SRS from baseline to 3 month after treatment to evaluate the effect of computer social interaction treatment on ASD children.
Autism Diagnostic Observation Schedule, ADOS | The baseline and 3 months after treatment
  The ADOS is a structured play session conducted by clinicians, with the total score combines the Social and Communication domain items, with high scores indicating severe symptoms. Change of the ADOS from baseline to 3 months after treatment to evaluate the effect of tablet computer social interaction treatment on ASD children.
Clinical Global Impression, CGI | The baseline and 3 months after treatment
  CGI is a scale used to assess the severity of the illness and the global improvement of the patient under intervention

OTHER OUTCOMES:
Head magnetic resonance imaging (MRI) | The baseline and 3 months after treatment
  Head MRI is used to detect the structure and function of the brain. Changes in the head MRI results of the subject before and after treatment.
Head functional Near infra-red spectroscopy (fNIRs) | The baseline and 3 months after treatment
  Head fNIRs is a non-invasive, non-ionizing method for measuring and imaging the functional hemodynamic response to brain activity. It measures changes in hemoglobin (Hb) concentrations within the brain by means of the characteristic absorption spectra of Hb in the near-infrared range. Changes in the head fNIRs results of the subject before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine